CLINICAL TRIAL: NCT00883636
Title: Cardiomyopathy in Steroid-resistant Nephrotic Syndrome: Impact of Focal Segmental Glomerulosclerosis
Status: Terminated | Type: Observational
Why Stopped: study stopped due to lack of activity
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: GCRC 0245; IRB# 08-163
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Focal Segmental Glomerulosclerosis; Nephrotic Syndrome; Steroid Resistant Nephrotic Syndrome; Chronic Kidney Disease
Keywords: Podocyte Protein; Podocyte Mutation
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrotic Syndrome; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Focal Segmental Glomerulosclerosis
  Interventions: Other: Cardiovascular Assessment; Other: Renal Assessment; Other: Genetic Evaluation
- Non-Focal Segmental Glomerulosclerosis
  Interventions: Other: Cardiovascular Assessment; Other: Renal Assessment; Other: Genetic Evaluation

INTERVENTIONS:
Other: Cardiovascular Assessment — Measure of BNP, and Pro-BNP Complete 2 Dimensional Echocardiogram with Doppler evaluation including determination of, Left Ventricular mass, Ejection fraction, Midwall fractional shortening, velocity of early and late diastolic transmitral flow, and measurement of E/A ratio, Ratio of end-systolic wall stress to rate corrected velocity of circumferential fiber shortening.
Other: Renal Assessment — Complete a metabolic panel, CMP. Calculation of glomerular filtration rate, GFR, measure of urinary total protein, albumin and creatinine excretion in a first morning urine sample, 24 hour blood pressure monitoring,
Other: Genetic Evaluation — All patients will undergo genetic screening for all known podocyte gene mutations.

SUMMARY:
The objective of this study is as follows:

* Perform genetic analysis to define the prevalence of each of the known gene mutations in an unselected cohort of patients with focal segmental glomerulosclerosis (FSGS)
* Perform a comprehensive assessment of cardiovascular status to determine the incidence of any cardiac abnormalities in patients with FSGS
* Determine if patients with mutations in specific proteins are more likely to have cardiovascular abnormalities
* Initiate long-term follow up in all patients to determine whether cardiac prognosis is related to any specific genetic abnormality

DETAILED DESCRIPTION:
Nephrotic Syndrome is a frequent cause of chronic kidney disease in children. Patients who are unresponsive to treatment with corticosteroids are further categorized as having steroid resistant nephrotic syndrome (SRNS). Renal biopsy in SRNS patients often reveal the histological lesion of focal segmental glomerulosclerosis (FSGS).

Genetic research has identified mutations in specific podocyte proteins, which may lead to the development of steroid resistant nephrotic syndrome. In addition to being expressed in the fetal adult kidney, human podocin mRNA is also expressed in the fetal heart tissue. Multiple case reports have described an association between cardiac abnormalities and familial FSGS. These findings suggest that this gene may be involved in the pathogenesis of cardiac abnormalities seen in this population.

The objectives of this study is to:

* Perform genetic analysis to define the prevalence of each of the known podocyte gene mutations in an unselected cohort of patients with FSGS
* Perform a comprehensive assessment of cardiovascular status to determine the incidence of any cardiac abnormalities in patients with FSGS
* Determine if patients with mutations in specific podocyte proteins are more likely to have cardiovascular abnormalities
* Initiate long-term follow up in all patients to determine whether cardiac prognosis is related to any specific genetic abnormality

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 21 years
* SRNS, defined as failure to achieve remission in proteinuria after 4-6 weeks of daily steroid therapy in accord with ISKDC guidelines
* GFR > 30 ml/min/1.73 m^2
* Renal disease diagnosed based on kidney biopsy

Exclusion Criteria:

* Secondary FSGS
* Prior renal transplantation
* Congenital extra-renal abnormalities
* Significant structural cardiac abnormalities
* pulmonary, hematologic, malignancy, or immune-related disease
* inability to maintain adequate follow-up

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Focal Segmental Glomerulosclerosis Patients and Non Focal Segmental Glomerulosclerosis SRNS patients
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Presence or Absence of any of the podocin gene mutations | baseline
  Presence or Absence of any of the podocin gene mutations
  1. podocin gene (NPHS2)
  2. CD2-associated protein (CD2AP)
  3. actinin-4 (ACTN4)
  4. Nephrotic syndrome steroid-resistant gene (SRN1)
  5. Wilms Tumor 1(WT1)
  6. Transient receptor potential cation channel, subfamily C, member 6 (TRPC6)
  7. Phospholipase C-E1 (PLCE-1)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Mensch, M.D., Principal Investigator — Northwell Health
Locations (1):
- Schneider Children's Hospital, New Hyde Park, New York, United States